CLINICAL TRIAL: NCT06489756
Title: Effect of Supplemental Oxygen Therapy (SOT) on Pulmonary Arterial Pressure in Highlanders With High Altitude Pulmonary Hypertension Permanently Living at >2500m
Brief Title: Highlanders With High Altitude Pulmonary Hypertension (HAPH), Pulmonary Arterial Pressure (PAP) Assessed at 3200m With and Without Supplemental Oxygen Therapy (SOT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HAPH_SOT_PAP
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; High Altitude; Supplemental Oxygen Therapy; Pulmonal Arterial Pressure
MeSH Terms: conditions — Pulmonary edema of mountaineers; Hypertension, Pulmonary; Hypoxia; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Each highlander with HAPH will perform a echocardiography with and without SOT according to a cross-over design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient air (Active Comparator): Highlanders with HAPH will perform the echocardiography on ambient air at 3200m
  Interventions: Other: Echocardiography
- 10 L/min SOT through face mask (Experimental): Supplemental oxygen therapy (SOT) at 10 L/min will be provided via face mask from oxygen concentrators
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Echocardiography will be performed according to clinical standards

SUMMARY:
The investigators aim to study the effect of SOT in highlanders with high altitude pulmonary hypertension (HAPH) who permanently live >2500m on pulmonary arterial pressure (PAP) assessed at 3200 m.

DETAILED DESCRIPTION:
Highlanders with HAPH diagnosed by echocardiography and defined by a RV/RA (Tricuspid Regurgitation Pressure Gradient) >30 mmHg will be recruited for this project. Highlanders permanently living at HA >2500 m will have echocardiografy to assess PAP near their living altitude in Aksay at 3200 m with and without 10L/min supplemental oxygen therapy (SOT) via face mask.

ELIGIBILITY:
Inclusion Criteria:

* Permanently living >2500 m
* HAPH diagnosed with a minimum RV/RA of 30 mmHg assessed by echocardiography at an altitude of 3200 m
* Written informed consent

Exclusion Criteria:

* Highlanders who cannot follow the study investigations,
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, heavy smoking >20 cigarettes/day or >20 pack-years.
* Coexistent unstable systemic hypertension or coronary artery disease that required adjustment of medication within the last 2 months
* Regular use of medication that affects control of breathing (benzodiazepines, opioids, acetazolamide)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Artery Pressure with SOT vs.ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Change in RV/RA in mmHg assessed by echocardiography with SOT compared to ambient air at 3200m

SECONDARY OUTCOMES:
Change in Cardiac Output with SOT vs. ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Change in cardiac output (l/min) assessed by echocardiography with SOT compared to ambient air at 3200m
Change in right to left heart diameter ratio with SOT vs.ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Change in right to left heart diameter ratio assessed by echocardiography with SOT compared to ambient air at 3200m
Change in tricuspid annular plane systolic excursion (TAPSE) with SOT vs.ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Change in tricuspid annular plane systolic excursion (TAPSE) with SOT compared to ambient air at 3200m
Change in right atrial area with SOT vs. ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Change in right atrial area by echocardiography with SOT compared to ambient air at 3200m
Change in right heart strain with SOT vs. ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Change in right heart strain by echocardiography with SOT compared to ambient air at 3200m
Change in pH by arterial blood gases with SOT vs. ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Changes in pH by arterial blood gases with SOT compared to ambient air at 3200m
Change in PaO2 by arterial blood gases with SOT vs. ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Changes in PaO2 by arterial blood gases with SOT compared to ambient air at 3200m
Change in PaCO2 by arterial blood gases with SOT vs. ambient air at 3200m | at 15 min of breathing ambient air or supplemental oxygen
  Changes in PaCO2 by arterial blood gases with SOT compared to ambient air at 3200m

CONTACTS AND LOCATIONS:
Overall Officials: Talant MA Sooronbaev, Prof. Dr., Principal Investigator — National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov; Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- Aksay Medical Center, Aksay Plateau, Naryn, Kyrgyzstan, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided